CLINICAL TRIAL: NCT05630794
Title: Phase 1 Trial of ONC201 for Chemoprevention in Colorectal Cancer
Brief Title: Testing for Safety and Colorectal Cancer Preventive Effects of ONC201
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2022-09737; NCI-2022-09737 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UMCC 2022.038 (Other: University of Michigan Rogel Cancer Center); UMI22-09-02 (Other: DCP); P30CA046592 (NIH); UG1CA242632 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2022-11-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Adenomatous Polyp; Colorectal Carcinoma; Familial Adenomatous Polyposis; Multiple Adenomatous Polyps
MeSH Terms: conditions — Colorectal Neoplasms; Adenomatous Polyposis Coli | interventions — Biopsy; Specimen Handling; Colonoscopy; TIC10 compound; Sigmoidoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (ONC201, biopsy, sigmoidoscopy, colonoscopy) (Experimental): Patients receive ONC201 PO QW or Q3W for 13 weeks. Patients also undergo collection of blood, tissue biopsy, and sigmoidoscopy/colonoscopy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Drug: Dordaviprone; Other: Questionnaire Administration; Procedure: Sigmoidoscopy

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Colonoscopy — Undergo colonoscopy
Drug: Dordaviprone — Given PO
  Other Names: Akt/ERK Inhibitor ONC201; ONC201; TIC10
Other: Questionnaire Administration — Ancillary studies
Procedure: Sigmoidoscopy — Undergo sigmoidoscopy
  Other Names: Proctosigmoidoscopy

SUMMARY:
The purpose of this phase I trial is to test the safety and cancer preventive effects of different doses of ONC201 in people with familial adenomatous polyposis (FAP) or a history of multiple polyps. People with familial adenomatous polyposis (FAP) or a history of multiple polyps are at higher than average risk of developing colorectal cancer. ONC201, now known as dordaviprone, is a drug that may stop cancer cells from growing. This drug has been shown in previous studies to cause cancer cell death but not harm normal cells. If successful, this study may help us develop a new option for colorectal cancer prevention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and toxicity of Akt/ERK Inhibitor ONC201 (ONC201) for the indication of cancer prevention in a healthy population of individuals who are at high risk (FAP and/or history of multiple adenomas [excluding hereditary nonpolyposis colorectal cancer (HNPCC)]) for recurrent colorectal adenomas.

SECONDARY OBJECTIVES:

I. To determine the dose(s) of ONC201 that yield(s) a statistically significant increase in human adenoma tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) expression.

II. To determine the dose(s) of ONC201 that yield(s) a statistically significant increase in normal human mucosa TRAIL expression.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of ONC201 on:

Ia. Cytokine/immune response profiles (with attention to interleukin [IL]-10, IL-17A, tumor necrosis factor [TNF]-alpha, IL-6, granzyme A, and perforin) in sera, normal colonic mucosa, and adenomas; Ib. Serum TRAIL concentration; Ic. Serum prolactin concentration; Id. Proliferation markers (Ki67), cell death markers (BCL2, Caspase 3), stemness markers (LGR5, CD44, CD133, ALDH), and natural killer (NK) cell infiltration in adenomas and in normal colonic mucosa; Ie. To evaluate for associations between observed toxicity and TRAIL expression; If. To establish organoids ex vivo and compare adenoma-derived organoid take rates between samples obtained prior to and following treatment.

OUTLINE: This is a dose-escalation study.

Patients receive ONC201 orally (PO) once weekly (QW) or once every 3 weeks (Q3W) for 13 weeks. Patients also undergo collection of blood, tissue biopsy, and sigmoidoscopy/colonoscopy throughout the study.

After completion of study treatment, patients are followed up at 21-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Be identified as high risk for recurrent colorectal adenomas, as defined by:

  * A diagnosis of FAP AND/OR
  * Findings of either > 5 small (less than 1 cm) adenomas OR >= 3 with at least one >= 10 mm on most recent colonoscopy performed in the past 5 years
* Be >= 18 years of age on day of signing informed consent
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum (glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase ([SGPT]) =< 1.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Participant is due to undergo a standard of care lower gastrointestinal (GI) colonoscopy for detection and removal of colorectal polyps. On this colonoscopy, participant is required to have:

  * Two (2) adenomatous polyps of at least five (5) mm in size
  * At least one (1) polyp within reach of a flexible sigmoidoscope (which will be retained in the colon or rectum and marked)
  * In addition to polypectomy, six (6) biopsies of normal colonic mucosa >= 1 cm from a collected polyp will also be collected
* Willing to undergo a second, research intent endoscopic procedure (either sigmoidoscopy or colonoscopy), approximately 12 weeks after initiating ONC201 treatment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Life expectancy of at least 5-years
* ONC201 is an imipridone agent with the potential for teratogenic or abortifacient effects. For this reason and because imipridones potential teratogenic effects are unknown, men and women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for four weeks after study treatment is completed. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should STOP the study medication and inform her study physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior history of hereditary nonpolyposis colorectal cancer (HNPCC), also known as Lynch syndrome
* Participants may not be currently receiving any other investigational agents or have received any investigational agents within the past four weeks
* Prior history of invasive colorectal cancer
* Prior invasive active neoplasm that is progressing or requires active treatment within 3 years from registration. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Participants with a history of prior invasive neoplasm diagnosed and treated greater than 3 years form registration may be considered with consultation of the primary investigator
* Prior history of exposure to cytotoxic chemotherapy or ONC201
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and women who are nursing are excluded from this study because ONC201 is an imipridone agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with ONC201, breastfeeding should be discontinued if the mother is treated with ONC201
* Concomitant use of strong CYP3A4/5 inducers/inhibitors. These agents must be discontinued at least 72-hours prior to beginning ONC201

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with unacceptable toxicity | Up to 35 days post last dose of ONC201
  Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Mean change in human adenoma tumor necrosis factor-related apoptosis-inducing ligand (TRAIL) expression in polyps induced by ONC201 | Baseline up to week 13 end of treatment
  The TRAIL expression in polyps obtained during pre-treatment colonoscopy and again during sigmoidoscopy after 12 weeks of treatment will be measured. The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.
Mean change in normal human mucosa TRAIL expression induced by ONC201 | Baseline up to week 13 end of treatment
  The TRAIL expression in polyps obtained during pre-treatment colonoscopy and again during sigmoidoscopy after 12 weeks of treatment will be measured. The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.

OTHER OUTCOMES:
Changes in mean cytokine/immune response levels (with attention to IL-10, IL-17A, TNFalpha, IL-6, granzyme A, and perforin) in sera, normal colonic mucosa, and adenomas between pre-, on-, and post-ONC201 treatment samples | Baseline up to week 13 end of treatment
  The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.
Changes in mean serum TRAIL concentrations in pre-, on-, and post-treatment samples obtained from participants treated with escalating doses of ONC201 | Baseline up to week 13 end of treatment
  The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.
Changes in mean serum prolactin concentrations in pre-, on-, and post-treatment samples obtained from participants treated with escalating doses of ONC201 | Baseline up to week 13 end of treatment
  The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.
Changes in Ki67, BCL2, Caspase 3, LGR5, CD44, CD133, and ALDH staining and NK cell infiltration in adenomas and in normal colonic mucosa obtained from participants prior to and following treatment with escalating doses of ONC201 | Baseline up to week 13 end of treatment
  The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.
Mean change in TRAIL expression between those who experience adverse events versus those who do not | Baseline up to week 13 end of treatment
  Will be compared qualitatively.
Adenoma-derived organoid take rates between samples obtained prior to and following treatment | Baseline up to week 13 end of treatment
  The mean difference in this change is compared between time points by means of a paired t-test. For skewed outcomes, the nonparametric Wilcoxon signed-rank test will be employed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Raufi, MD, Principal Investigator — Brown University and Rhode Island Hospital
Locations (5):
- United States (5):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm